CLINICAL TRIAL: NCT06403631
Title: Supporting Mental Health in Daily Life After the Diagnosis of Multiple Sclerosis: the Role of Flow Experience and Mindfulness
Brief Title: Supporting Mental Health in Daily Life After the Diagnosis of Multiple Sclerosis
Acronym: MindFlowMS
Status: Recruiting | Type: Observational
Sponsor: Marta Bassi (Other)
Collaborators: Italian Multiple Sclerosis Foundation (Other); Università Vita-Salute San Raffaele (Other); Azienda Ospedaliera Sant'Anna (Other); San Luigi Gonzaga Hospital (Other); University of Florence (Other); University of Bari (Other); University of Cagliari (Other); Azienda Ospedaliera San Camillo Forlanini (Other); University of Catania (Other)
Responsible Party: Sponsor-Investigator, Marta Bassi, Associate Professor, University of Milan
Organization: University of Milan (Other)
Other Study IDs: 2022/R-Multi/020
Record Dates: First submitted 2024-04-25; First posted 2024-05-08 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational — Data will be gathered longitudinally from participants newly diagnosed with multiple sclerosis. Participants will fill in online questionnaires measuring flow, mindfulness, positive mental health, anxiety and depression. The questionnaires, including both scaled and open-ended questions, will be proposed at the project start (T1) and 6 months later (T2).

SUMMARY:
The overall goal of this observational study is to learn about the psychological resources of mindfulness and flow experience available to persons newly diagnosed with multiple sclerosis (MS). The primary study aim will be to analyze the relation of flow and mindfulness with mental health among individuals who received an MS diagnosis within the last year. Secondary aims will be to analyze the daily activities preferentially associated with flow, and to evaluate possible changes in daily flow retrieval. Participants will answer questionnaires measuring flow, mindfulness, positive mental health, anxiety and depression at project start and 6 months later.

DETAILED DESCRIPTION:
The period following Multiple Sclerosis (MS) diagnosis is extremely important to identify and mobilize psychological resources that can support mental health, help cope with challenges, and lead to disease acceptance. Capitalizing on previous studies attesting to the crucial role of attentional skills in disease adjustment, the overall goal of this project is to jointly investigate flow experience and mindfulness as potential resources supporting mental health among newly diagnosed persons. While mindfulness has been widely investigated in relation to MS, flow has been rarely explored. Both constructs are rewarding mental states involving focused attention on the present moment and perceived control over the situation. Yet, they also present relevant differences. Mindfulness is characterized by reflective awareness, while flow by loss of selfconsciousness. Mindfulness can generate initial heightened unpleasant feelings, and its cultivation requires constant practice; instead, flow does not require intensive training and it is reported in association with ordinary daily situations and activities. In light of these differences, it may be suitable to promote flow, or a combination of flow and mindfulness, at the initial stages of MS, as newly diagnosed persons require immediate psychological support and need to find a sense of continuity in life. The primary study aim will be to analyze the relation of flow and mindfulness with mental health among individuals who received an MS diagnosis within the last year.

Secondary aims will be to analyze the daily activities preferentially associated with flow, and to evaluate possible changes in daily flow retrieval. Data will be gathered longitudinally from participants recruited in MS centers across Italy. Participants will fill in online questionnaires measuring flow, mindfulness, positive mental health, anxiety and depression. The questionnaires, including both scaled and open-ended questions, will be proposed at the project start (T1) and 6 months later (T2). Hierarchical regressions and qualitative analyses will be conducted to assess study aims. Both flow and mindfulness are expected to independently contribute to participants' mental health. However, considering its usual occurrence in daily contexts, flow is expected to provide a more relevant contribution than mindfulness, and to play a moderating role in the relation between mindfulness and mental health. The investigators also expect that participants will primarily retrieve flow in productive and leisure activities, and that fewer participants would find flow occasions in their daily life after the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50
* clinically-definite MS diagnosed (with McDonald's revised criteria) within the previous 12 months
* steroid treatment for at least 1 month
* written informed consent

Exclusion Criteria:

* neurological disorders other than MS
* psychiatric disorders
* severe physical impairment (EDSS=>8)
* pregnancy
* current or previous attendance in Mindfulness Based Interventions or Acceptance and Commitment Therapy
* severe cognitive impairment in comprehension, attention and execution of inferential-logical operations which could interfere with the ability to fill in questionnaires (equivalent scores 0-1 at Progressive Raven Matrices; score <11.3 at the visual comprehension of sentences subtest of the Aphasia Neuropsychological Test; score <37.9 at Symbol Digit Modalities Test; and score <93.1 at the Brief Test of Intelligence)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Outpatients of Neurological Units
Sampling Method: Non-Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Positive mental health (Mental Health Continuum Short Form) | The questionnaires will be administered at T1 (within 12 months from diagnosis disclosure) and at T2 (after 6 months)
  Mental Health Continuum Short Form, min-max sum values: 0-70, higher scores indicating higher mental health
Anxiety (subscale of the Hospital Anxiety and Depression Scale) | The questionnaires will be administered at T1 (within 12 months from diagnosis disclosure) and at T2 (after 6 months)
  Subscale of the Hospital Anxiety and Depression Scale, min-max sum values: 0-21, higher scores indicating higher anxiety levels
Depression (subscale of the Hospital Anxiety and Depression Scale) | The questionnaires will be administered at T1 (within 12 months from diagnosis disclosure) and at T2 (after 6 months)
  Subscale of the Hospital Anxiety and Depression Scale, min-max sum values: 0-21, higher scores indicating higher depression levels

SECONDARY OUTCOMES:
Flow-related activities (Flow Questionnaire) | The questions will be administered at T1 (within 12 months from diagnosis disclosure) and at T2 (after 6 months)
  Flow Questionnaire: open-ended questions on activities associated with flow experience
Flow occurrence (Flow Questionnaire) | The questionnaire will be administered at T1 (within 12 months from diagnosis disclosure) and at T2 (after 6 months)
  Flow Questionnaire: dummy variable for flow presence (1) vs. absence (0)

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - University of Bari, Bari
  - University of Cagliari, Cagliari
  - University of Catania, Catania
  - Azienda Ospedaliera Sant'Anna, Como
  - University of Florence, Florence
  - Università Vita-Salute San Raffaele, Milan
  - San Luigi Gonzaga Hospital, Orbassano
  - Azienda Ospedaliera San Camillo Forlanini, Roma

IPD SHARING:
Plan to Share IPD: No